CLINICAL TRIAL: NCT06643494
Title: Alleviating Androgen Deprivation Therapy (ADT) + External Beam Radiation (EBR) Treatment Side Effects in Prostate Cancer Patients
Brief Title: Elimination of Prostate Cancer Treatment Side Effects Using a Nutraceutical
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PPI currently unable to continue.
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RLP051624.
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study consists of a single group of subjects included in the study design, in which all subjects receive a single intervention, N-111, and the outcomes are assessed over time.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both the active compactor and the placebo will be in unlabeled foil packets. The contents will be the same weight and color.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- N-111 (Active Comparator): Nutraceutical N-111 in conjunction with ADT + EBR will be given in this arm, once per day with breakfast.
  Interventions: Dietary Supplement: N-111
- Placebo (Placebo Comparator): A placebo that is inert but appears to look the same as the active comparator in conjunction with ADT + EBR, given once per day with breakfast.
  Interventions: Other: Placebo
- Control (No Intervention): The control group will proceed with the ADT + EBR treatment without taking the active compactor or the placebo.

INTERVENTIONS:
Dietary Supplement: N-111 — A combination of Acetogenins
  Arms: N-111
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Does nutraceutical N-111 lower the number of side effects occurring during ADT + External Beam Radiation (EBR) prostate cancer treatment?

DETAILED DESCRIPTION:
Researchers will compare nutraceutical N-111 to a placebo (a look-alike substance that contains no active ingredients) and control group to see if N-111 works to alleviate side effects of prostate cancer treatment.

Participants will:

Take N-111 or a placebo by mouth every day for the duration of the ADT + EBR therapy. Fill out the self-evaluation reporting form weekly during EBR therapy and every three months during ADT therapy to assess their symptoms or lack of symptoms.

The patients will see a physician once a week during the EBR therapy and once every three months for the duration of the ADT therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male undergoing treatment for prostate cancer with ADT + EBR.

Exclusion Criteria:

* Everyone else

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 100 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Self-reporting | Weekly for the duration of EBR (6 weeks). Monthly for the duration of ADT (2 years).
  Self-reporting symptom severity and number of symptoms. The scoring is from 1 (no issue) to 10 (severe), across 14 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Jeppsen, MD, Study Chair — Optimal Health Research
Locations (1):
- Optimal Health Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No